CLINICAL TRIAL: NCT07263022
Title: Cognitive Strategies in Early Psychosis 2
Acronym: COSTEP 2
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY00025575; P50MH119569 (NIH)
Record Dates: First submitted 2025-08-25; First posted 2025-12-04 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Psychosis; Schizophrenia Disorder; Schizoaffective Disorder; Major Depressive Disorder With Psychotic Features; Bipolar Disorder With Psychotic Features; Psychosis NOS; Schizophreniform Disorder; Psychotic Disorder; Cognition
Keywords: Cognition; Decision Making; fMRI; Psychosis spectrum disorders
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Mental Disorders | interventions — Modafinil

STUDY DESIGN:
Intervention Model Description: Each participant will take a single dose of each drug 2 times. There will be 6 different orders of administration (e.g., A>B>C, A>C>B).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm 1: Modafinil > d-serine > placebo (Experimental): Participants will take single doses three study medications in the following order: modafinil (200mg); d-serine (100mg/kg); and placebo. All medications will be taken 2 times (A>B>C>A>B>C).
  (Note: This order is not necessarily reflective of the actual randomization schedule used in the protocol, as the procedure is double-blinded)
  Interventions: Drug: Modafinil; Drug: D-serine solution; Drug: Placebo
- Arm 2: Modafinil > placebo > d-serine (Experimental): Participants will take single doses of three study medications in the following order: modafinil (200mg); placebo; and d-serine (100mg/kg). All medications will be taken 2 times (A>B>C>A>B>C).
  (Note: This order is not necessarily reflective of the actual randomization schedule used in the protocol, as the procedure is double-blinded)
  Interventions: Drug: Modafinil; Drug: D-serine solution; Drug: Placebo
- Arm 3: D-serine > modafinil > placebo (Experimental): Participants will take single doses of three study medications in the following order: d-serine (100mg/kg); modafinil (100mg); and placebo. All medications will be taken 2 times (A>B>C>A>B>C).
  (Note: This order is not necessarily reflective of the actual randomization schedule used in the protocol, as the procedure is double-blinded)
  Interventions: Drug: Modafinil; Drug: D-serine solution; Drug: Placebo
- Arm 4: D-serine > placebo > modafinil (Experimental): Participants will take single doses of three study medications in the following order: d-serine (100mg/kg); placebo; and modafinil (100mg). All medications will be taken 2 times (A>B>C>A>B>C).
  (Note: This order is not necessarily reflective of the actual randomization schedule used in the protocol, as the procedure is double-blinded)
  Interventions: Drug: Modafinil; Drug: D-serine solution; Drug: Placebo
- Arm 5: Placebo > modafinil > d-serine (Experimental): Participants will take single doses of three study medications in the following order: placebo; modafinil (100 mg); and d-serine (100 mg/kg). All medications will be taken 2 times (A>B>C>A>B>C).
  (Note: This order is not necessarily reflective of the actual randomization schedule used in the protocol, as the procedure is double-blinded)
  Interventions: Drug: Modafinil; Drug: D-serine solution; Drug: Placebo
- Arm 6: Placebo > d-serine > modafinil (Experimental): Participants will take single doses of three study medications in the following order: placebo; d-serine (100 mg/kg); and modafinil (100mg). All medications will be taken 2 times (A>B>C>A>B>C).
  (Note: This order is not necessarily reflective of the actual randomization schedule used in the protocol, as the procedure is double-blinded)
  Interventions: Drug: Modafinil; Drug: D-serine solution; Drug: Placebo

INTERVENTIONS:
Drug: Modafinil — Single dose of modafinil capsule, 100 mg. Participants will also receive an oral placebo solution to maintain the blind.
Drug: D-serine solution — Single dose of oral solution of d-serine, 100 mg/kg. Participants will also receive a placebo capsule to maintain the blind.
Drug: Placebo — Single dose of oral placebo, in both capsule and oral solution

SUMMARY:
The goal of this clinical trial is to learn more about decision making in psychosis spectrum disorders, like schizophrenia. Participants will be people who have had symptoms of a psychosis spectrum disorder start within the last five years. The investigators will study how two study agents change decision making in people with psychosis, by asking participants to complete some brain games on the computer before and after taking the study agents. The investigators hope to improve our understanding of psychosis to help people in the future. The main research questions are:

* Does a single dose of modafinil change how people with psychosis play the brain games?
* Does a single dose of d-serine change how people with psychosis play the brain games?
* Does a single dose of modafinil change brain activity?
* Does a single dose of d-serine change brain activity?

Participants will:

* Complete an interview and self-report questionnaires.
* Complete safety screening activities, like a blood draw, a urine drug test, and an alcohol breathalyzer test.
* Complete functional Magnetic Resonance Imaging (fMRI) scans. fMRI uses magnets to take pictures of the brain. There will be six scanning appointments in the study, with two scans each. Appointments will be about a month apart.
* Take a single dose of a study agent during each scanning appointment. The study agent will be taken after the first fMRI. There are three study agents in total: modafinil, d-serine, and a placebo. Each participant will take each study agent twice during the study.
* Play brain games on a computer that measure decision making, thinking, and problem solving skills

DETAILED DESCRIPTION:
Participants will be asked to complete ten appointments in this study: An intake appointment, 6 functional Magnetic Resonance Imaging (fMRI) appointments, and 3 clinical interview appointments. In addition, there will be 3 brief clinical check ins, and 6 phone call check ins after fMRI appointments.

Intake Appointment:

The first appointment is the Intake appointment. This visit will take between 1.75-2.75 hours, depending on how many study tasks are needed. Participants in this study may have participated in a sister study, called "State Representation in Early Psychosis 2 (STEP 2)." If so, they will not need to complete many of the intake questionnaires, and it is expected to take about 100 minutes for them to complete this appointment. If they did not participate in STEP 2, participants will need to complete the full intake battery.

During the interview, the investigators will ask questions about a participant's medical and psychiatric history, and current and past mental health symptoms. They will collect demographics, as well as information on the person's social life and quality of life. Participants will also provide a blood sample for clinical safety screening. The investigators will collect one 3mL tube, which is less than 2/3 of a teaspoon. If pregnancy is a physical possibility, they will also collect a urine sample for pregnancy testing.

fMRI Appointments: The second appointment is an fMRI + study agent appointment. Participants will come in person to the University of Minnesota Center for Magnetic Resonance Research. This visit will take about 7-7.5 hours.

First, the investigators will complete safety screening measures. This will include:

* A screening questionnaire to make sure the participant can enter the fMRI machine safely
* A blood pressure reading.
* A vision test.
* A breathalyzer to test for the presence of alcohol.
* A urine drug test to screen for the presence of substances.
* If pregnancy is a physical possibility, a urine pregnancy test will be required.

After screening measures are successfully completed, participants will complete the brain games on a computer. Afterwards, the participant will enter the fMRI machine. The very first fMRI scan will last 2 hours, as the investigators will get additional pictures for the structure of the brain before the scan that measures brain activity.

After this, the participant will take a single dose of the study agent. Neither the participant nor the study team will know which study agent the participant is taking. They will be randomly assigned to one of six schedules (for example, one participant will have A > B > C, and another will have A > C > B, and so on). The participant will be provided with a meal while the study agent metabolizes. Afterwards, the investigators will monitor the participant's vital signs and ask whether they are experiencing any adverse effects.

After the observation period is completed, the participant will complete a second fMRI scan. This scan will last 90 minutes. Afterwards, they will play the same brain games on the computer. The investigators will take another vital sign measurement and ask about adverse effects.

The following day, the investigators will contact the participant via phone to ask whether they experienced any adverse effects after leaving the study appointment. This call should last about 5 minutes.

The remaining 5 fMRI visits will be the same, except that the first scan of the day will be only 90 minutes long. fMRI appointments will be scheduled approximately one month apart.

Clinical Interview Appointments:

Between fMRIs 1 and 2, 3 and 4, and 5 and 6, the investigators will interview participants to ask questions about their current mental health symptoms, their quality of life, and their social life. Participants will also complete self-report questionnaires which cover the same topics. These appointments will take about 90 minutes. The appointment can be completed in person at the University of Minnesota or remotely via Zoom.

Between fMRIs 2 and 3, and 4 and 5, participants will be asked a brief series of questions about their recent mental health symptoms. This will be a remote visit conducted via Zoom or by phone. These calls should take about 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 35
* Onset of a psychosis spectrum illness (schizophrenia, schizoaffective disorder, schizophreniform disorder, psychosis NOS, bipolar disorder with psychosis, or major depressive disorder with psychosis) within 5 years of enrollment
* Estimated IQ of 70 or above
* Proficient at English as determined through interactions with the study team
* No change in psychiatric medication within a week of enrollment or MRI study visits
* No clinically significant change in any medications for at least 1 month prior to study participation or MRI study visits, as determined by PI/Co-Is

  * Participants may have minor adjustments in medication doses in the past 30 days, per PI discretion, but may not have had major increases or decreases in doses, or additions or removal of medication within the past 30 days.
  * Participants are to have no changes to medications in the past 7 days before drug administration (i.e., must have been on a stable dose for at least 7 days prior to receiving the study drug).

Exclusion Criteria:

Medical Criteria:

* Presence of the following medical concerns as determined by the study PI:

  * Major neurological disorder
  * History of a clinically significant head injury with or without prolonged unconsciousness
  * Any major medical condition that, in the opinion of the PI, would impede participation in the study or would put the participant at additional risk by participating
* History of any of the following as reported by the participant:

  * Renal impairment, injury, or disease
  * Hepatic impairment, injury, or disease
  * Myocardial infarction or heart disease, or endorsement of history of or of cardiac symptoms at intake:

    * Dyspnea
    * Palpitations
    * Orthopnea
    * Pedal oedema
    * Significant dizziness
    * Syncope
    * Claudication
  * Low white blood cell count, or is diagnosed with leukopenia, neutropenia, or agranulocytosis
* Presence of unmanaged hypertension (>140/90) or elevated resting heart rate (>100 bpm)
* Abnormal clinical laboratory values:

  * uACR > 30 mg/g
  * creatinine level >0.95 mg/dL
  * AST or ALT > 50 U/L
  * Bilirubin > 1.2 mg/dL
  * Total Protein < 6 g/dL
* Taking a medication or supplement that has a major drug interaction with any study drugs (e.g., ketamine, MAOIs, clomipramine, diazepam, propranolol, warfarin)
* Allergies to study drugs
* Is pregnant, planning to become pregnant, or is breastfeeding
* Cannot pass the visual acuity test
* Cannot pass the CMRR Subject Safety Screen due to MRI contraindications

Mental health criteria:

* Meets criteria for a severe substance or alcohol use disorder within 3 months of enrollment
* Lifetime history of a stimulant use disorder
* Current manic episode as determined by the MINI
* History of psychiatric hospitalization within 3 months of enrollment
* Meets criteria for clinical risk of suicidal behavior, as defined by:

  * Clinician judgment
  * A suicide attempt within 3 months of enrollment
  * Active suicidal ideation at screening or baseline, as indicated by the C-SSRS Screener
  * Previous intent to act on suicidal ideation with a specific plan and/or preparatory acts within 3 months of enrollment, as indicated by the C-SSRS Screener
* Symptom severity scores in the severe (6) or extremely severe (7) range on the BPRS for the following items: suicidality, disorientation, bizarre behavior, excitement, elevated mood
* Any other psychiatric symptoms or conditions that, in the opinion of the PI, would impede participation in the study or put the participant at additional risk by participating

Other criteria:

* Unable or unwilling to provide informed consent
* Unable to demonstrate adequate decisional capacity, in the judgment of the consenting study staff member, to make a choice about participating in the research study
* Current guardianship
* Is under civil commitment or under a stay of civil commitment
* Illiteracy
* Has engaged in significant cognitive training, in the opinion of the PI, in the last year

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Test My Brain - Digit Symbol Coding | Baseline
  A computerized cognitive assessment measuring processing speed. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Digit Symbol Coding | Day 7 (fMRI 1)
  A computerized cognitive assessment measuring processing speed. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Digit Symbol Coding | Day 36 (fMRI 2)
  A computerized cognitive assessment measuring processing speed. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Digit Symbol Coding | Day 63 (fMRI 3)
  A computerized cognitive assessment measuring processing speed. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Digit Symbol Coding | Day 91 (fMRI 4)
  A computerized cognitive assessment measuring processing speed. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Digit Symbol Coding | Day 119 (fMRI 5)
  A computerized cognitive assessment measuring processing speed. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Digit Symbol Coding | Day 147 (fMRI 6)
  A computerized cognitive assessment measuring processing speed. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Verbal Paired Associates Memory | Baseline
  A computerized cognitive assessment measuring verbal memory. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Verbal Paired Associates Memory | Day 7 (fMRI 1)
  A computerized cognitive assessment measuring verbal memory. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Verbal Paired Associates Memory | Day 36 (fMRI 2)
  A computerized cognitive assessment measuring verbal memory. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Verbal Paired Associates Memory | Day 63 (fMRI 3)
  A computerized cognitive assessment measuring verbal memory. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Verbal Paired Associates Memory | Day 91 (fMRI 4)
  A computerized cognitive assessment measuring verbal memory. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Verbal Paired Associates Memory | Day 119 (fMRI 5)
  A computerized cognitive assessment measuring verbal memory. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Verbal Paired Associates Memory | Day 147 (fMRI 6)
  A computerized cognitive assessment measuring verbal memory. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Matrix Reasoning | Baseline
  A computerized cognitive assessment measuring problem solving. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Matrix Reasoning | Day 7 (fMRI 1)
  A computerized cognitive assessment measuring problem solving. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Matrix Reasoning | Day 36 (fMRI 2)
  A computerized cognitive assessment measuring problem solving. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Matrix Reasoning | Day 63 (fMRI 3)
  A computerized cognitive assessment measuring problem solving. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Matrix Reasoning | Day 91 (fMRI 4)
  A computerized cognitive assessment measuring problem solving. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Matrix Reasoning | Day 119 (fMRI 5)
  A computerized cognitive assessment measuring problem solving. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Matrix Reasoning | Day 147 (fMRI 6)
  A computerized cognitive assessment measuring problem solving. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Multiracial Emotion Identification | Baseline
  A computerized cognitive assessment measuring social cognition and emotion recognition skills. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Multiracial Emotion Identification | Day 7 (fMRI 1)
  A computerized cognitive assessment measuring social cognition and emotion recognition skills. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Multiracial Emotion Identification | Day 36 (fMRI 2)
  A computerized cognitive assessment measuring social cognition and emotion recognition skills. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Multiracial Emotion Identification | Day 63 (fMRI 3)
  A computerized cognitive assessment measuring social cognition and emotion recognition skills. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Multiracial Emotion Identification | Day 91 (fMRI 4)
  A computerized cognitive assessment measuring social cognition and emotion recognition skills. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Multiracial Emotion Identification | Day 119 (fMRI 5)
  A computerized cognitive assessment measuring social cognition and emotion recognition skills. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Multiracial Emotion Identification | Day 147 (fMRI 6)
  A computerized cognitive assessment measuring social cognition and emotion recognition skills. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Resting-state functional connectivity | Day 7 (fMRI 1)
  Resting state connectivity in the brain is measured with fMRI. The primary outcome will be changes in resting-state functional connectivity before and after study agent administration
Resting-state functional connectivity | Day 36 (fMRI 2)
  Resting state connectivity in the brain is measured with fMRI. The primary outcome will be changes in resting-state functional connectivity before and after study agent administration
Resting-state functional connectivity | Day 63 (fMRI 3)
  Resting state connectivity in the brain is measured with fMRI. The primary outcome will be changes in resting-state functional connectivity before and after study agent administration
Resting-state functional connectivity | Day 91 (fMRI 4)
  Resting state connectivity in the brain is measured with fMRI. The primary outcome will be changes in resting-state functional connectivity before and after study agent administration
Resting-state functional connectivity | Day 119 (fMRI 5)
  Resting state connectivity in the brain is measured with fMRI. The primary outcome will be changes in resting-state functional connectivity before and after study agent administration
Resting-state functional connectivity | Day 147 (fMRI 6)
  Resting state connectivity in the brain is measured with fMRI. The primary outcome will be changes in resting-state functional connectivity before and after study agent administration
Dot Pattern Expectancy variation (TOPX) task performance | Day 7 (fMRI 1)
  The TOPX task consists of a series of pattern sequences. One pattern is designated the "A" cue, and another the "X" cue, which requires one response (AX, 60-70% of trials, e.g. respond with the left button), while other sequences require a different response (AY or BX, 12-15% of trials each, or BY, 6-10% of trials, e.g. respond with the right button). Given the strong expectation that X's evokes a valid response, BX trials place demands on the fidelity (stability, memory) of the "B" cue state representation to overcome this tendency. Performance is assessed based on accuracy and response time. The primary outcome will be differences in task performance before and after modafinil administration.
Dot Pattern Expectancy variation (TOPX) task performance | Day 36 (fMRI 2)
  The TOPX task consists of a series of pattern sequences. One pattern is designated the "A" cue, and another the "X" cue, which requires one response (AX, 60-70% of trials, e.g. respond with the left button), while other sequences require a different response (AY or BX, 12-15% of trials each, or BY, 6-10% of trials, e.g. respond with the right button). Given the strong expectation that X's evokes a valid response, BX trials place demands on the fidelity (stability, memory) of the "B" cue state representation to overcome this tendency. Performance is assessed based on accuracy and response time. The primary outcome will be differences in task performance before and after modafinil administration.
Dot Pattern Expectancy variation (TOPX) task performance | Day 63 (fMRI 3)
  The TOPX task consists of a series of pattern sequences. One pattern is designated the "A" cue, and another the "X" cue, which requires one response (AX, 60-70% of trials, e.g. respond with the left button), while other sequences require a different response (AY or BX, 12-15% of trials each, or BY, 6-10% of trials, e.g. respond with the right button). Given the strong expectation that X's evokes a valid response, BX trials place demands on the fidelity (stability, memory) of the "B" cue state representation to overcome this tendency. Performance is assessed based on accuracy and response time. The primary outcome will be differences in task performance before and after modafinil administration.
Dot Pattern Expectancy variation (TOPX) task performance | Day 91 (fMRI 4)
  The TOPX task consists of a series of pattern sequences. One pattern is designated the "A" cue, and another the "X" cue, which requires one response (AX, 60-70% of trials, e.g. respond with the left button), while other sequences require a different response (AY or BX, 12-15% of trials each, or BY, 6-10% of trials, e.g. respond with the right button). Given the strong expectation that X's evokes a valid response, BX trials place demands on the fidelity (stability, memory) of the "B" cue state representation to overcome this tendency. Performance is assessed based on accuracy and response time. The primary outcome will be differences in task performance before and after modafinil administration.
Dot Pattern Expectancy variation (TOPX) task performance | Day 119 (fMRI 5)
  The TOPX task consists of a series of pattern sequences. One pattern is designated the "A" cue, and another the "X" cue, which requires one response (AX, 60-70% of trials, e.g. respond with the left button), while other sequences require a different response (AY or BX, 12-15% of trials each, or BY, 6-10% of trials, e.g. respond with the right button). Given the strong expectation that X's evokes a valid response, BX trials place demands on the fidelity (stability, memory) of the "B" cue state representation to overcome this tendency. Performance is assessed based on accuracy and response time. The primary outcome will be differences in task performance before and after modafinil administration.
Dot Pattern Expectancy variation (TOPX) task performance | Day 147 (fMRI 6)
  The TOPX task consists of a series of pattern sequences. One pattern is designated the "A" cue, and another the "X" cue, which requires one response (AX, 60-70% of trials, e.g. respond with the left button), while other sequences require a different response (AY or BX, 12-15% of trials each, or BY, 6-10% of trials, e.g. respond with the right button). Given the strong expectation that X's evokes a valid response, BX trials place demands on the fidelity (stability, memory) of the "B" cue state representation to overcome this tendency. Performance is assessed based on accuracy and response time. The primary outcome will be differences in task performance before and after modafinil administration.
Translational Bandit Task (TBT) Performance | Day 7 (fMRI 1)
  This is a task variant that uses choice options (neutral images) that are rewarded probabilistically. The rewarded stimulus with the highest reward is changed over time. State learning associated with staying or switching stimuli too quickly (lose-switching) can be evaluated. Performance is assessed based on accuracy, response time, and behavior of reward seeking. The primary outcome will be differences in task performance before and after modafinil administration.
Translational Bandit Task (TBT) Performance | Day 36 (fMRI 2)
  This is a task variant that uses choice options (neutral images) that are rewarded probabilistically. The rewarded stimulus with the highest reward is changed over time. State learning associated with staying or switching stimuli too quickly (lose-switching) can be evaluated. Performance is assessed based on accuracy, response time, and behavior of reward seeking. The primary outcome will be differences in task performance before and after modafinil administration.
Translational Bandit Task (TBT) Performance | Day 63 (fMRI 3)
  This is a task variant that uses choice options (neutral images) that are rewarded probabilistically. The rewarded stimulus with the highest reward is changed over time. State learning associated with staying or switching stimuli too quickly (lose-switching) can be evaluated. Performance is assessed based on accuracy, response time, and behavior of reward seeking. The primary outcome will be differences in task performance before and after modafinil administration.
Translational Bandit Task (TBT) Performance | Day 91 (fMRI 4)
  This is a task variant that uses choice options (neutral images) that are rewarded probabilistically. The rewarded stimulus with the highest reward is changed over time. State learning associated with staying or switching stimuli too quickly (lose-switching) can be evaluated. Performance is assessed based on accuracy, response time, and behavior of reward seeking. The primary outcome will be differences in task performance before and after modafinil administration.
Translational Bandit Task (TBT) Performance | Day 119 (fMRI 5)
  This is a task variant that uses choice options (neutral images) that are rewarded probabilistically. The rewarded stimulus with the highest reward is changed over time. State learning associated with staying or switching stimuli too quickly (lose-switching) can be evaluated. Performance is assessed based on accuracy, response time, and behavior of reward seeking. The primary outcome will be differences in task performance before and after modafinil administration.
Translational Bandit Task (TBT) Performance | Day 147 (fMRI 6)
  This is a task variant that uses choice options (neutral images) that are rewarded probabilistically. The rewarded stimulus with the highest reward is changed over time. State learning associated with staying or switching stimuli too quickly (lose-switching) can be evaluated. Performance is assessed based on accuracy, response time, and behavior of reward seeking. The primary outcome will be differences in task performance before and after modafinil administration.

SECONDARY OUTCOMES:
Brief Psychiatric Rating Scale (BPRS) - Global Score | Baseline
  Clinician-administered rating scale to assess psychiatric symptoms such as depression, anxiety, hallucinations, and unusual behavior. Scores on individual items range from 1 (not present) to 7 (extremely severe); global scores range from 24 to 168
Brief Psychiatric Rating Scale (BPRS) - Global Score | Day 21 (Clinical A)
  Clinician-administered rating scale to assess psychiatric symptoms such as depression, anxiety, hallucinations, and unusual behavior. Scores on individual items range from 1 (not present) to 7 (extremely severe); global scores range from 24 to 168
Brief Psychiatric Rating Scale (BPRS) - Global Score | Day 49 (Brief Clinical B)
  Clinician-administered rating scale to assess psychiatric symptoms such as depression, anxiety, hallucinations, and unusual behavior. Scores on individual items range from 1 (not present) to 7 (extremely severe); global scores range from 24 to 168
Brief Psychiatric Rating Scale (BPRS) - Global Score | Day 77 (Clinical C)
  Clinician-administered rating scale to assess psychiatric symptoms such as depression, anxiety, hallucinations, and unusual behavior. Scores on individual items range from 1 (not present) to 7 (extremely severe); global scores range from 24 to 168
Brief Psychiatric Rating Scale (BPRS) - Global Score | Day 105 (Brief Clinical D)
  Clinician-administered rating scale to assess psychiatric symptoms such as depression, anxiety, hallucinations, and unusual behavior. Scores on individual items range from 1 (not present) to 7 (extremely severe); global scores range from 24 to 168
Brief Psychiatric Rating Scale (BPRS) - Global Score | Day 133 (Clinical E)
  Clinician-administered rating scale to assess psychiatric symptoms such as depression, anxiety, hallucinations, and unusual behavior. Scores on individual items range from 1 (not present) to 7 (extremely severe); global scores range from 24 to 168
Scale for Assessment of Negative Symptoms/Scale for Assessment of Positive Symptoms (SANS/SAPS) - Global score | Day 21 (Clinical A)
  The SANS (25 items) and SAPS (34 items) are clinician-administered scales that assess negative and positive symptoms of schizophrenia. Individual items are rated from 0 (symptoms not present) to 5 (Marked symptoms); global scores range from 0 to 295.
Scale for Assessment of Negative Symptoms/Scale for Assessment of Positive Symptoms (SANS/SAPS) - Global score | Day 77 (Clinical C)
  The SANS (25 items) and SAPS (34 items) are clinician-administered scales that assess negative and positive symptoms of schizophrenia. Individual items are rated from 0 (symptoms not present) to 5 (Marked symptoms); global scores range from 0 to 295.
Scale for Assessment of Negative Symptoms/Scale for Assessment of Positive Symptoms (SANS/SAPS) - Global score | Day 133 (Clinical E)
  The SANS (25 items) and SAPS (34 items) are clinician-administered scales that assess negative and positive symptoms of schizophrenia. Individual items are rated from 0 (symptoms not present) to 5 (Marked symptoms); global scores range from 0 to 295.

OTHER OUTCOMES:
Abbreviated Quality of Life Scale (aQLS) - Global Score | Day 21 (Clinical A)
  Clinician-administered rating scale to assess functioning in schizophrenia. Individual items range from 0 (virtually absent) to 6 (Little or no deficit); global scores range from 0 to 54.
Abbreviated Quality of Life Scale (aQLS) - Global Score | Day 77 (Clinical C)
  Clinician-administered rating scale to assess functioning in schizophrenia. Individual items range from 0 (virtually absent) to 6 (Little or no deficit); global scores range from 0 to 54.
Abbreviated Quality of Life Scale (aQLS) - Global Score | Day 133 (Clinical E)
  Clinician-administered rating scale to assess functioning in schizophrenia. Individual items range from 0 (virtually absent) to 6 (Little or no deficit); global scores range from 0 to 54.
Global Functioning - Social Scale (GFS) | Clinical A
  Clinician-administered rating scale to assess social functioning. Scores range from 1 (extreme social isolation) to 10 (Superior social/interpersonal functioning)
Global Functioning - Social Scale (GFS) | Day 77 (Clinical C)
  Clinician-administered rating scale to assess social functioning. Scores range from 1 (extreme social isolation) to 10 (Superior social/interpersonal functioning)
Global Functioning - Social Scale (GFS) | Day 133 (Clinical E)
  Clinician-administered rating scale to assess social functioning. Scores range from 1 (extreme social isolation) to 10 (Superior social/interpersonal functioning)
Global Functioning - Role Scale (GFR) | Day 21 (Clinical A)
  Clinician-administered rating scale to assess occupational functioning. Scores range from 1 (Extreme role dysfunction) to 10 (Superior role functioning)
Global Functioning - Role Scale (GFR) | Day 77 (Clinical C)
  Clinician-administered rating scale to assess occupational functioning. Scores range from 1 (Extreme role dysfunction) to 10 (Superior role functioning)
Global Functioning - Role Scale (GFR) | Day 133 (Clinical E)
  Clinician-administered rating scale to assess occupational functioning. Scores range from 1 (Extreme role dysfunction) to 10 (Superior role functioning)

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Vinogradov, MD, Principal Investigator — University of Minnesota Department of Psychiatry and Behavioral Sciences; Caroline Demro, Ph.D., Principal Investigator — University of Minnesota Department of Psychiatry and Behavioral Sciences

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with the National Institutes of Mental Health Data Archive (collection ID pending).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared 1 year following study completion. There is no end date for data sharing.
Access Criteria: Users who register with the NIMH Data Archive will be able to access the data.